CLINICAL TRIAL: NCT02875925
Title: Pharmacist-provided Medication Management in Medicare-ACO Patients Taking Medications Associated With Medication-related Hospitalization or Emergency Visits in the Elderly
Brief Title: Outcomes Study of MTM in a Medicare ACO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthEast Care System (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSSMMTM1
Record Dates: First submitted 2016-08-15; First posted 2016-08-23 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2017-06

CONDITIONS: Pain; Hypoglycemia
Keywords: blood coagulation
MeSH Terms: conditions — Pain; Hypoglycemia; Thrombosis | interventions — Medication Therapy Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MTM (Experimental): Patients will receive MTM at an individualized frequency for 1 year.
  Interventions: Other: MTM
- Control (No Intervention): Patients enrolled in the control group will not experience any change in their medical care.

INTERVENTIONS:
Other: MTM — Medication management is a process that ensures each patient's medications are assessed to determine the appropriateness, effectiveness, safety, and convenience of each medication for the patient. Medication management is fully integrated with the care team. Pharmacists provide this service to identify, prevent, and resolve drug therapy problems improve outcomes.
  Other Names: Medication Management
  Arms: MTM

SUMMARY:
This is a non-randomized, prospective, quasi-experimental study designed to assess the impact of pharmacist-provided medication management on total cost of care and clinical outcomes (ie, hospitalizations, emergency department visits) in a real-world clinical practice.

DETAILED DESCRIPTION:
Medication Management (MTM)

Medication management is defined as the standard of care that ensures each patient's medications, including prescription, over-the-counter, herbal products, vitamins, and supplements, are individually assessed to determine the following:

* Appropriateness of each medication for the patient
* Effectiveness for the patient's medical conditions
* Safety given the patient's co-morbidities and other medications
* Convenience to be taken by the patient as intended

Medication management services are delivered to an individual patient and are fully integrated with the health care team to achieve coordinated and consistent patient care. Pharmacists provide this service using a standardized method to comprehensively review each patient's medications. This systematic process is designed to identify, prevent, and resolve drug therapy problems and to aid in attainment of a patient's therapy goals. Medication management services include an individualized care plan that tracks progress on the intended goals of therapy with appropriate follow-up to determine actual patient outcomes. Pharmacists aim to emphasize the care experience for patients, achieve better medication-related quality measures, and reduce the cost of care.

Patients who are enrolled in the MTM group will have an initial MTM visit, which will last approximately 60 minutes. In this visit, the patient and the pharmacist will discuss all medications (prescription, over-the-counter, and herbal) that the patient is taking. Medications will be evaluated for indication, efficacy, safety and convenience. The pharmacist and patient and other care team members will participate in shared decision in an effort to optimize patient clinical outcomes and medication experience. Patients will continue to work with their primary care provider and other care team members. Patients will continue to meet with the pharmacist on an individualized basis for 1 year to optimize the patients' medications based on individual needs.

Patients enrolled in the control group will not experience any change in their medical care on account of being enrolled in the control group. They will continue to work with their primary care provider and other care team members.

ELIGIBILITY:
Inclusion Criteria:

* MSSP patient, attributed to Community Health Network
* Receive primary care at HealthEast as demonstrated by having > 2 outpatient visits at one of HealthEast's primary care clinics in the 3 years prior to enrollment.
* Currently taking > 1 medication from the following therapeutic classes: antiplatelet/anticoagulant, hypoglycemic (oral or insulin), opioid analgesic
* Willingness of subject to work with a MTM pharmacist for medication management throughout the 12 month study period.
* Provided written informed consent

Exclusion Criteria:

* Currently receiving their primary care at a non-HealthEast clinic
* Inpatient status at Bethesda Hospital within last 12 months
* Currently receiving hospice care
* In the opinion of the investigator, have any kind of disorder that may compromise the ability of the subject to provide written informed consent

Min Age: 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 77 (Actual)
Dates: Start 2015-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Hospitalization Rates | 12 months
Emergency Department Visits | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Wallace, PharmD, MS, Principal Investigator — HealthEast Care System
Locations (1):
- HealthEast Care System, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes